CLINICAL TRIAL: NCT05991804
Title: Upper Limb Spinal Cord Stimulation for Rehabilitation Enhancement
Acronym: Up-Stim
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 319893
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries
Keywords: Rehabilitation; Transcutaneous spinal cord stimulation; Upper limb
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham transcutaneous spinal cord stimulation (placebo) added to inpatient rehabilitation (Active Comparator): Standard inpatient rehabilitation received at the Royal National Orthopaedic Hospital NHS Trust
  Interventions: Other: Sham transcutaneous spinal cord stimulation (placebo) added to inpatient rehabilitation
- Transcutaneous spinal cord stimulation added to inpatient rehabilitation (Experimental): Transcutaneous spinal cord stimulation added to standard inpatient rehabilitation, targetting the upper limbs, received at the Royal National Orthopaedic Hospital NHS Trust
  Interventions: Other: Transcutaneous spinal cord stimulation added to inpatient rehabilitation

INTERVENTIONS:
Other: Transcutaneous spinal cord stimulation added to inpatient rehabilitation — Non-invasive electrical stimulation delivered over the spine, targetting movement of the upper limbs
  Arms: Transcutaneous spinal cord stimulation added to inpatient rehabilitation
Other: Sham transcutaneous spinal cord stimulation (placebo) added to inpatient rehabilitation — Sham transcutaneous spinal cord stimulation (placebo) added to Standard inpatient rehabilitation given at the Royal National Orthopaedic Hospital NHS Trust
  Arms: Sham transcutaneous spinal cord stimulation (placebo) added to inpatient rehabilitation

SUMMARY:
In the United Kingdom, there are more than 1000 new cases of spinal cord injury (SCI) each year, with around half of these injuries affecting the cervical spine. People who have reduced function and control affecting their upper limbs may have difficulty carrying out activities of daily living (ADLs), significantly affecting their independence. Recovering even partial upper limb function is a top priority among tetraplegics.

Regaining voluntary function in the upper limb can have a huge impact on quality of life. Using TSCS in the upper limb for acute SCI can benefit patients early in their rehabilitation, and may reduce the number of patients with problematic spasticity at discharge. Transcutaneous spinal cord stimulation (TSCS) may provide a low-cost method of improving function and spasticity in this cohort.

The aim of this feasibility study is to assess and compare the impact of adding TSCS to the standard rehabilitation of inpatients with acute SCI, compared to a sham (placebo) TSCS intervention added to standard rehabilitation, in an effort to enhance upper limb control and function.

DETAILED DESCRIPTION:
Recruitment:

Participants will be recruited from the Royal National Orthopaedic Hospital. A member of our research team will contact participants after they have received this information sheet to discuss participation in the study and answer any questions. People who would like to take part in the study will be asked to attend an initial session to see if they are able to tolerate non-invasive SCS.

Intervention:

Eligible participants will then be randomised either into the intervention group, where they will receive TSCS or sham TSCS in addition to their regular inpatient rehabilitation. We are using this trial design to assess whether adding TSCS to regular inpatient rehabilitation enhances recovery and voluntary function in this participant cohort, and to test that there is not a placebo effect.

For both the sham and intervention groups, we will carry out regular assessments. Some of these assessments will be part of standard care as an inpatient at the RNOH, and others will be additional. Please see the outcome measures for further information about these assessments.

Follow-up:

When participants have finished their inpatient rehabilitation at the RNOH, we will carry out a semi-structured interview, where we will ask about participants' experience on this study. Interviews may take place in person, over the phone, or over video call (e.g. Microsoft Teams or Zoom).

Participants will then be invited to two Follow-up Assessments at the RNOH, where all outcome measures will be repeated. Follow-up 1 will be done once the participant is 6-months post-injury, and Follow-up 2 will be done at 1-year post-injury. If the participant is already 6-months post-injury at discharge, then Follow-up 1 will occur at 1-month post-discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18
2. Recent spinal cord injury (inpatient at the RNOH)
3. Spinal cord injury level C1-C8
4. AIS A-D
5. Willing and able to provide informed consent

Exclusion Criteria:

1. Women who are pregnant, planning pregnancy or breastfeeding
2. Those who have a cardiac pacemaker
3. Active device at stimulating electrode site
4. Any other musculoskeletal diagnosis affecting the upper limbs
5. Spinal malignancy
6. Spinal cord injury due to cancerous growth
7. Auto-immune disorder
8. Ongoing infection
9. Uncontrolled autonomic dysreflexia
10. Complex regional pain syndrome
11. Neurological degenerative diseases
12. Peripheral nerve damage affecting the upper limbs
13. Taking part in a conflicting research study
14. People who are unable to tolerate TSCS during their first session

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2028-04-16 (Estimated); Study Completion 2028-04-16 (Estimated)

PRIMARY OUTCOMES:
Change in International Standards of Neurological Classification for SCI (ISNC-SCI). | 30 minutes
  This is a is a clinician-administered scale used to classify the severity (completeness) of injury in individuals with SCI.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | 20 minutes
  This is a is a clinician-administered scale used to classify spasticity
Range of Motion (ROM) | 20 minutes
  This is a is a clinician-administered scale used to classify the angles that can be achieved at each joint of the arm
Electromyography (EMG) assessments | 90 minutes
  This will be assessed by researchers, and classifies the amount of muscle activity occurring during movements of the arms and hands.
Individual goal planning | 20 minutes
  This is planned between the participant and their therapist, and defines what is important to the participant to gain from their rehabilitation
Spinal Cord Independence Measure (SCIM) | 30 minutes
  This is a self-assessed outcome which asks the rater about 3 areas of function: self-care (feeding, grooming, bathing, and dressing), respiration and sphincter management, and mobility
Tetraplegic upper limb activity questionnaire (TUAQ) | 30 minutes
  This is a self-assessed questionnaire which is a self-assessment of hand and arm function
International SCI data sets quality of life basic data set (SCI-QoL) | 15 minutes
  This is a self-administered short questionnaire which assesses quality of life
Semi-structured interview | 60 minutes
  Participants will be asked to speak freely about their experience on this project and any recommendations they have for the team for future studies

CONTACTS AND LOCATIONS:
Overall Officials: Lynsey Duffell, PhD, Principal Investigator — University College, London
Locations (1):
- Royal National Orthopaedic Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
As the study is only 6 participants IPD will be provided in study publications.